CLINICAL TRIAL: NCT01872520
Title: Post-marketing Safety Surveillance of the Injection of DanShenDuoFenSuanYan (the Injection of Depsides Salts From Salvia Miltiorrhiza): A Real World Study
Brief Title: Post-marketing Safety Surveillance of the Injection of DanShenDuoFenSuanYan A Real World Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Shanghai Greenvalley Pharmaceutical Co., Ltd. (Industry); Peking University (Other)
Responsible Party: Principal Investigator, Suodi ZHAI, Suodi ZHAI, Department of Pharmacy, Peking University Third Hospital, Peking University Third Hospital
Other Study IDs: PekingUTH-Pharmacy-001
Record Dates: First submitted 2013-04-13; First posted 2013-06-07 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Adverse Drug Reaction
Keywords: the Injection of DanShenDuoFenSuanYan; Magnesium Lithospermate B; Safety; Real World Study
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- the Injection of DanShenDuoFenSuanYan: Patient who use the Injection of DanShenDuoFenSuanYan

SUMMARY:
Magnesium Lithospermate B, the main constituent of the Injection of DanShenDuoFenSuanYan (the Injection of Depsides Salts From Salvia Miltiorrhiza), is the active ingredient of Salvia Miltiorrhiza. This study record clinical use of The injection of DanShenDuoFenSuanYan in the real world, and observe the adverse drug reactions/ adverse drug events during treatment.

DETAILED DESCRIPTION:
As a traditional chinese medicine, the Injection of DanShenDuoFenSuanYan (the Injection of Depsides Salts From Salvia Miltiorrhiza) was approved by State Food and Drug Administration of China in May,2005. This cardiovascular drug is one of the few Traditional Chinese Medicine pharmaceuticals where the active ingredients have been identified in the molecular levels. In its 8 years marketing in China, there is no serious adverse drug reactions.

In this study, clinical pharmacists in selected hospitals will record the clinical use and the adverse drug reactions/ adverse drug events of this injection.

This real world study for the Injection of DanShenDuoFenSuanYan with 30400 patients will be conducted from June.2012 to May.2014.

ELIGIBILITY:
Inclusion Criteria:

* Patients who use the Injection of DanShenDuoFenSuanYan in 30 hospitals in china(including the inpatient and the outpatient(only in some hospitals which can get the information)).

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who use the Injection of DanShenDuoFenSuanYan in 30 hospitals in china(including the inpatient and the outpatient(only in some hospitals which can get the information))
Sampling Method: Non-Probability Sample
Enrollment: 30180 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The incidence of IDSDFSY induced adverse drug reaction | 3 years
The rare adverse drug reactions to the IDSDFSY | 3 years

SECONDARY OUTCOMES:
The manifestation, treatment and outcomes of the ADRs | 3 years
  To describe manifestation, treatment and outcomes of the ADRs.
The risk factors of the ADRs | 3 years
  To examine the risk factors of the ADRs.
The patients' characteristics who are prescribed IDSDFSY | 3 years
  To describe the patients' characteristics who are prescribed IDSDFSY.
The prescribing pattern of IDSDFSY in real world clinical practice | 3 years
  To characterize the prescribing pattern of IDSDFSY in real world clinical practice.
Off-label use of IDSDFSY | 3 years
  To describe and evaluate the off-label use of IDSDFSY.

CONTACTS AND LOCATIONS:
Overall Officials: Suodi ZHAI, B.S., Study Chair — Peking University Third Hospital
Locations (36):
- China (36):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Guang'anmen Hospital affiliatied to China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking university third hospital, Beijing, Beijing Municipality
  - The Military General Hospital of Beijing PLA, Beijing, Beijing Municipality
  - The General Hospital of People's Liberation Army(301 hospital), Beijing, Beijing Municipality
  - First Hospital Of Qinhuangdao, Qinhuangdao, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Hebei General Hospital, Shijiazhuang, Hebei
  - Wuhan Hospital of Traditional Chinese Medicine, Wuhan, Hubei
  - Wuhan Asia Heart Hospital, Wuhan, Hubei
  - Wuhan Integrated TCM and Western Medicine Hospital, Wuhan, Hubei
  - Hubei Provincial Hospital of TCM, Wuhan, Hubei
  - Zhangjiagang Hospital Of Traditional Chinese Medicine, Zhangjiagang, Jiangsu
  - Weinan Central Hospital, Weinan, Shaanxi
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing hospital, Xi'an, Shaanxi
  - Shaanxi Province Hospital of Traditional Chinese Medicine, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Yanan University Affiliated Hospital, Yan’an, Shaanxi
  - Shanghai Huangpu District Central Hospital, Shanghai, Shanghai Municipality
  - Shuguang Hospital Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Longhua Hospital Shanghai University of TCM, Shanghai, Shanghai Municipality
  - Minhang District Central Hospital, Shanghai, Shanghai Municipality
  - Central Hospital Of Qingpu District, Shanghai, Shanghai, Shanghai Municipality
  - Sichuan 2nd Hospital Of TCM, Chengdu, Sichuan
  - Hospital Of Chengdu Office Of People's Government of Tibetan Autonomous Region (Hospital.C.T.), Chengdu, Sichuan
  - Affiliated Hospital of Chengdu University, Chengdu, Sichuan
  - AVIC 363 Hospital, Chengdu, Sichuan
  - China S.C.H.J. Hospital Of TCM, Hejiang, Sichuan
  - The First Affiliated Hospital of the Medical College, Shihezi University, Shihezi, Xinjiang
  - The Fifth Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Traditional Chinese Medicine Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - Chest Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Derived] Yan YY, Yang YH, Wang WW, Pan YT, Zhan SY, Sun MY, Zhang H, Zhai SD. Post-Marketing Safety Surveillance of the Salvia Miltiorrhiza Depside Salt for Infusion: A Real World Study. PLoS One. 2017 Jan 26;12(1):e0170182. doi: 10.1371/journal.pone.0170182. eCollection 2017. PMID 28125608